CLINICAL TRIAL: NCT05652985
Title: Effect of Inter-professional Collaboration Training Program on Nurses' Collegial Solidarity and Knowledge Sharing: A Randomized Controlled Trial
Brief Title: Effect of Inter-professional Collaboration Training Program on Nurses' Collegial Solidarity and Knowledge Sharing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Port Said University (Other)
Responsible Party: Principal Investigator, Heba Emad Elgazar, lecture of nursing administraion, Port Said University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NUR (6/11/2022) (19)
Record Dates: First submitted 2022-11-29; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Nurses Behaviors
Keywords: Inter-professional Collaboration; Collegial Solidarity; Knowledge Sharing

STUDY DESIGN:
Intervention Model Description: open-label, two-arm Randomized Control Trail (RCT)
Masking Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): Inter-professional Collaboration Training
  Interventions: Behavioral: Inter-professional Collaboration Training
- control group (No Intervention): Regarding the control group, the participants will receive no training

INTERVENTIONS:
Behavioral: Inter-professional Collaboration Training — the participated nurses will receive session about Inter-professional Collaboration followed by activity which can boost Inter-professional Collaboration
  Arms: interventional group

SUMMARY:
Effect of Inter-professional Collaboration Training Program on Nurses' Collegial Solidarity and Knowledge Sharing

DETAILED DESCRIPTION:
the study aims to evulate the effectiveness of inter-professional collaboration training program on nurses' collegial solidarity and knowledge sharing

Hypotheses:

H1: Nurses participating in the inter-professional collaboration training program will report, post intervention, high level of inter-professional collaboration behaviors compared with those nurse nurses in control group.

H2: Nurses participating in the inter-professional collaboration training program will report, post intervention, high level of collegial solidarity compared with those nurse nurses in control group H3: Nurses participating in the inter-professional collaboration training program will report, post intervention, high level of knowledge sharing compared with those nurse nurses in control group this is RCT study among nurses work in EL-Salam hospital, port said, Egypt

ELIGIBILITY:
Inclusion Criteria:

* licensed nurses who worked in direct contact with patients in their services
* had at least six month of experience in the nursing profession,
* agreed to participate in the study

Exclusion Criteria:

* participating in any intervention program within the last 12 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Inter-professional collaboration of nurses | 3 monthes
  measuring changes occure in inter-professional collaboration behaviours after applied . inter-professional collaboration training. the researchers will use Inter-professional collaboration competency scale developed by Yamamoto et al. (2014) in an English language and will be translated to Arabic language by the researcher. It consisted of 40 items designed to evaluate interprofessional collaboration competency in six factors: respecting patients (5 items); team management skills, (5 items); fulfilling one's role as a professional, (4 items); attitudes and beliefs as a professional, (6 items); attitudes that improve team cohesion (4 items); and taken to achieve the team's goal. (6 items). using a Likert scale from one to five where one equals "disagree" and five equals "agree". Higher scores indicate stronger interprofessional collaboration.

SECONDARY OUTCOMES:
Colleage solidatory among nurses | 3 months
  measuring changes occure in colleage solidatory after applied inter-professional collaboration training. Colleague Solidarity Scale Developed by Uslusoy and Alpar (2013). will be used. It consisted of 23 items designed to evaluate collegial solidarity in three factors: emotional solidarity (9 items); academic solidarity, (9 items); and negative opinions about solidarity. (5 items). sing a Likert scale from one to five where one equals "never" and five equals "always". Subscale scores of the colleague solidarity scale are calculated by summing the scores of the constituent items of each subscale; higher scores indicate stronger collegial solidarity.
knoweledge sharing | 3 months
  the researchers will use Knowledge Sharing Readiness scale to measure change occuring in knoweledge sharining behaviours after program application. This tool adopted from Ridder and deVries (2006) consisting of 16 items. donating (8items) and collecting (8items). Scoring system: Nurses' responses will be measured on a five point Likert scale ranging from "one= strongly disagree, two =disagree, three =uncertain, four = agree, and five = strongly agree".

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication will be shared to open data repository.
Supporting Information: Study Protocol
Time Frame: the data will be available after publishing the trail (expected in 2023)
Access Criteria: Open access